CLINICAL TRIAL: NCT04084366
Title: A Phase 1/2, Open-Label, Dose-Escalation and Cohort-Expansion Study Evaluating the Safety, Pharmacokinetics, and Therapeutic Activity of OBI-999 in Patients With Advanced Solid Tumors
Brief Title: Phase 1/2 Study of OBI-999 in Patients With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Has not shown its expected therapeutic potential for the enrolled patients in this trial
Sponsor: OBI Pharma, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: OBI-999-001
Record Dates: First submitted 2019-09-05; First posted 2019-09-10 (Actual); Results first posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Locally Advanced Solid Tumor
Keywords: antibody drug conjugate (ADC)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- OBI-999 Escalation phase (Experimental): Part A: Five cohorts at escalating dose levels 0.4, 0.8, 1.2, 1.6 and 2.0 mg/kg (capping calculations at a maximum at 100 kg) of OBI-999 liquid form via IV infusion to establish maximum tolerated dose (MTD) and Recommended phase 2 dose (RP2D).
  Interventions: Drug: OBI-999
- OBI-999 Expansion Phase (Experimental): Part B: Five cohorts of patients at RP2D of OBI-999 liquid form, as determined from Part A, via IV infusion.
  Interventions: Drug: OBI-999

INTERVENTIONS:
Drug: OBI-999 — For the dose-escalation phase, OBI-999 will be administered on Day 1 of each 21-day cycle, for up to 35 cycles.
  Arms: OBI-999 Escalation phase
Drug: OBI-999 — For the dose-expansion phase, OBI-999 will be administered on Day 1 of each 21-day cycle, for up to 35 cycles.
  Arms: OBI-999 Expansion Phase

SUMMARY:
The purpose of this study is to establish the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) of OBI-999 as monotherapy, and to characterize the safety and preliminary clinical activity profile of the RP2D of OBI-999 in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients, 18 years of age or older at the time of consent.
2. Provide written informed consent prior to performing any study related procedure.
3. Histologically or cytologically confirmed patients with advanced solid tumors.
4. Patients must have been treated with established standard-of-care therapy, or physicians have determined that such established therapy is not sufficiently efficacious, or patients have declined to receive standard-of-care therapy. In the latter case, the informed consent must state the effective therapies the patient is declining.
5. Measurable disease (i.e., at least one measurable lesion per RECIST 1.1)
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
7. Adequate organ function defined as:

   a. Hepatic:

   i. Serum ALT ≤3 × upper limit of normal (ULN), ≤5 × ULN in the presence of liver metastases

   ii. Serum AST ≤3 × ULN, ≤5 × ULN in presence of liver metastases

   iii.Serum bilirubin ≤1.5 × ULN (unless due to Gilbert's syndrome or hemolysis)

   b. Renal:

   i. Creatinine clearance >50 mL/minute using Cockcroft Gault equation

   c. Hematologic:

   i. Absolute neutrophil count ≥1,500/µL

   ii. Platelets ≥100,000/µL

   iii. Hemoglobin ≥8 g/dL
8. Patient is willing and able to comply with all protocol required assessments, visits, and procedures, including a pretreatment tumor biopsy. Archival tumor biopsies are acceptable at baseline.
9. Females of childbearing potential must have negative serum pregnancy test prior to starting study therapy, and agree to use a reliable form of contraceptive during the study treatment period and for at least 120 days following the last dose of study drug.

   Patient not of childbearing potential (i.e., permanently sterilized, postmenopausal) can be included in study. Postmenopausal is defined as 12 months with no menses without an alternative medical cause.

   Male patients must agree to use an adequate method of contraception during the study treatment period and for at least 120 days following the last dose of study drug.
10. Cannot be breast feeding.
11. Patients with human immunodeficiency virus (HIV) infection are eligible if CD4+ T cell counts ≥ 350 cells/uL; patients on antiretroviral therapy (ART) should be on an established dose for at least 4 weeks and have an HIV viral load less than 400 copies/mL prior to enrollment.
12. Patients with serological evidence of chronic hepatitis B virus (HBV) infection are eligible if they have an HBV viral load below the limit of quantification with or without concurrent viral suppressive therapy.
13. Patients with a history of hepatitis C virus (HCV) infection should have completed curative antiviral treatment and have a viral load below the limit of quantification.
14. Patients in Part B (Cohort-Expansion) must have documented Globo H H score of at least 100 from a qualified laboratory IHC assay in one of the sponsor-selected tumor types to be enrolled in the respective cohort:

    * Cohort 1: Pancreatic cancer
    * Cohort 2: Esophageal cancer
    * Cohort 3: Gastric cancer
    * Cohort 4: Colorectal cancer
    * Cohort 5: Basket (any solid tumor type other than those included in Cohorts 1 through 4).

Exclusion Criteria:

1. Less than 3 weeks from prior cytotoxic chemotherapy or radiation therapy; and less than 5 half-lives or 3 weeks, whichever is shorter, from prior biologic therapies, prior to the first dose of OBI 999.
2. Has undergone a major surgical procedure (as defined by the Investigator) or significant traumatic injury within 28 days prior to the first dose of OBI 999.
3. Sensory or motor neuropathy of Grade 2 or greater.
4. Patients with a history of solid organ transplant.
5. Unresolved toxicities from prior anticancer therapy, defined as having not resolved to Grade 0 or 1 (using NCI CTCAE version 5.0), except for alopecia and laboratory values listed in the inclusion criteria.
6. Receipt of any prior therapy targeting Globo H.
7. Known hypersensitivity to OBI 999 or its excipients.
8. Has known untreated central nervous system metastases. Patients with treated brain metastases are eligible if there is no evidence of progression for at least 4 weeks after CNS-directed treatment, as ascertained by clinical examination and brain imaging (magnetic resonance imaging [MRI] or computed tomography [CT]) during the screening period.
9. Has significant clinical cardiac abnormality (e.g., clinical heart failure or unstable angina)
10. Any medical co morbidity that is life threatening or, in the opinion of the Investigator, renders the patient unsuitable for participation in a clinical trial due to possible noncompliance, would place the patient at an unacceptable risk and/or potential to affect interpretation of results of the study.
11. Is receiving any concurrent prohibited medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2019-11-25 (Actual); Primary Completion 2023-10-27 (Actual); Study Completion 2023-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Apostolia Tsimberidou, MD, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (4):
- United States (4):
  - Scripps MD Anderson Cancer Center, La Jolla, California
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - West Cancer Center, Germantown, Tennessee
  - University of Texas MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tsimberidou AM, Vo HH, Beck J, Shia CS, Hsu P, Pearce TE. First-in-Human Study of OBI-999, a Globo H-Targeting Antibody-Drug Conjugate, in Patients With Advanced Solid Tumors. JCO Precis Oncol. 2023 Jan;7:e2200496. doi: 10.1200/PO.22.00496. PMID 36701651

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A, Dose Escalation - OBI-999 0.4 mg/kg: OBI-999 0.4 mg/kg was administered as an IV infusion on Day 1 of each 21-day cycle
- Part A, Dose Escalation - OBI-999 0.8 mg/kg: OBI-999 0.8 mg/kg was administered as an IV infusion on Day 1 of each 21-day cycle
- Part A, Dose Escalation - OBI-999 1.2 mg/kg; Part B, Cohort Expansion - Cohort 1, Pancreatic; Part B, Cohort Expansion - Cohort 2, Colorectal Cancer; Part B, Cohort Expansion - Cohort 3, Basket (Any Other Solid Tumor Other Than Cohorts 1 and 2): OBI-999 1.2 mg/kg was administered as an IV infusion on Day 1 of each 21-day cycle
- Part A, Dose Escalation - OBI-999 1.6 mg/kg: OBI-999 1.6 mg/kg was administered as an IV infusion on Day 1 of each 21-day cycle
Period: Overall Study
Arm/Group | Part A, Dose Escalation - OBI-999 0.4 mg/kg | Part A, Dose Escalation - OBI-999 0.8 mg/kg | Part A, Dose Escalation - OBI-999 1.2 mg/kg | Part A, Dose Escalation - OBI-999 1.6 mg/kg | Part B, Cohort Expansion - Cohort 1, Pancreatic | Part B, Cohort Expansion - Cohort 2, Colorectal Cancer | Part B, Cohort Expansion - Cohort 3, Basket (Any Other Solid Tumor Other Than Cohorts 1 and 2)
Started | 3 | 3 | 6 | 3 | 11 | 10 | 8
Completed | 0 | 0 | 0 | 0 | 1 | 0 | 2
Not Completed | 3 | 3 | 6 | 3 | 10 | 10 | 6

BASELINE CHARACTERISTICS:
Population: The safety population consisted of all enrolled subjects who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A, Dose Escalation - OBI-999 0.4 mg/kg | Part A, Dose Escalation - OBI-999 0.8 mg/kg | Part A, Dose Escalation - OBI-999 1.2 mg/kg | Part A, Dose Escalation - OBI-999 1.6 mg/kg | Part B, Cohort Expansion - Cohort 1, Pancreatic | Part B, Cohort Expansion - Cohort 2, Colorectal Cancer | Part B, Cohort Expansion - Cohort 3, Basket (Any Other Solid Tumor Other Than Cohorts 1 and 2) | Total
Number analyzed (Participants) | 3 | 3 | 6 | 3 | 11 | 10 | 8 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.7 (16.44) | 70.3 (5.13) | 55.2 (8.47) | 54.7 (18.9) | 62.1 (11.48) | 59.6 (10.66) | 62.9 (8.15) | 60.2 (11.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 3 | 2 | 5 | 5 | 4 | 20
  Male | 2 | 3 | 3 | 1 | 6 | 5 | 4 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 3
  Not Hispanic or Latino | 3 | 2 | 2 | 3 | 11 | 7 | 8 | 36
  Unknown or Not Reported | 0 | 0 | 3 | 0 | 0 | 2 | 0 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race (custom): American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Race (custom): Asian | 0 | 0 | 0 | 0 | 4 | 2 | 3 | 9
  Race (custom): Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Race (custom): Black or African American | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 3
  Race (custom): White | 3 | 2 | 4 | 1 | 7 | 5 | 5 | 27
  Race (custom): Other | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 3
  Race (custom): More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Race (custom): Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 6 | 3 | 7 | 9 | 6 | 37
  Taiwan | 0 | 0 | 0 | 0 | 4 | 1 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) (CR+PR)
Description: Assessment of OBI-999 clinical benefit rate for dose escalation and cohort expansion phases of the OBI 999-001 study.
Time Frame: Every 6 weeks (±7 days) for first 3 months, then every 9 weeks (±7 days) until discontinuation of study treatment, disease progression, death, or initiation of further cancer therapy, or for up to 35 cycles (approximately 2 years.), whichever occurs first
Population: The efficacy population consists of all patients who are enrolled, have received at least 1 dose of study drug, and had at least one follow-up tumor assessment scan.
Measure: Number (95% Confidence Interval); unit: % of participants
Arm/Group | Part A, Dose Escalation - OBI-999 0.4 mg/kg | Part A, Dose Escalation - OBI-999 0.8 mg/kg | Part A, Dose Escalation - OBI-999 1.2 mg/kg | Part A, Dose Escalation - OBI-999 1.6 mg/kg | Part B, Cohort Expansion - Cohort 1, Pancreatic | Part B, Cohort Expansion - Cohort 2, Colorectal Cancer | Part B, Cohort Expansion - Cohort 3, Basket (Any Other Solid Tumor Other Than Cohorts 1 and 2)
Number analyzed (Participants) | 3 | 3 | 6 | 3 | 7 | 8 | 8
% of participants | 0 [0 to 70.8] | 0 [0 to 70.8] | 0 [0 to 45.9] | 0 [0 to 70.8] | 0 [0 to 41] | 0 [0 to 36.9] | 0 [0 to 36.9]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for up to approximately 2 years after first dose
Description: Treatment-emergent adverse events (TEAEs) in Parts A or B experienced by ≥5% of total subjects in Part A and Part B. TEAEs are presented by decreasing incidence for the total of subjects in Part A and Part B
Arm/Group | Part A, Dose Escalation - OBI-999 0.4 mg/kg | Part A, Dose Escalation - OBI-999 0.8 mg/kg | Part A, Dose Escalation - OBI-999 1.2 mg/kg | Part A, Dose Escalation - OBI-999 1.6 mg/kg | Part B, Cohort Expansion - Cohort 1, Pancreatic | Part B, Cohort Expansion - Cohort 2, Colorectal Cancer | Part B, Cohort Expansion - Cohort 3, Basket (Any Other Solid Tumor Other Than Cohorts 1 and 2)
All-Cause Mortality (participants affected / at risk) | 1/3 | 1/3 | 0/6 | 1/3 | 3/11 | 1/10 | 1/8
Serious Adverse Events (participants affected / at risk) | 2/3 | 1/3 | 2/6 | 3/3 | 8/11 | 2/10 | 0/8
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 5/6 | 3/3 | 10/11 | 10/10 | 7/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A, Dose Escalation - OBI-999 0.4 mg/kg (N=3) | Part A, Dose Escalation - OBI-999 0.8 mg/kg (N=3) | Part A, Dose Escalation - OBI-999 1.2 mg/kg (N=6) | Part A, Dose Escalation - OBI-999 1.6 mg/kg (N=3) | Part B, Cohort Expansion - Cohort 1, Pancreatic (N=11) | Part B, Cohort Expansion - Cohort 2, Colorectal Cancer (N=10) | Part B, Cohort Expansion - Cohort 3, Basket (Any Other Solid Tumor Other Than Cohorts 1 and 2) (N=8)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Klebsiella sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Biliary obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A, Dose Escalation - OBI-999 0.4 mg/kg (N=3) | Part A, Dose Escalation - OBI-999 0.8 mg/kg (N=3) | Part A, Dose Escalation - OBI-999 1.2 mg/kg (N=6) | Part A, Dose Escalation - OBI-999 1.6 mg/kg (N=3) | Part B, Cohort Expansion - Cohort 1, Pancreatic (N=11) | Part B, Cohort Expansion - Cohort 2, Colorectal Cancer (N=10) | Part B, Cohort Expansion - Cohort 3, Basket (Any Other Solid Tumor Other Than Cohorts 1 and 2) (N=8)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 | 2 (3) | 1 (1) | 2 (2) | 0 | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 0 | 4 (4) | 2 (2) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 | 1 (1) | 1 (2) | 0 (0) | 1 (2) | 3 (4) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 0 | 0 | 0 | 2 (3) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 | 0 | 2 (2) | 0 | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 | 1 (1) | 1 (1) | 0 | 0 | 2 (2) | 2 (2)
Fatigue (General disorders) | 2 (2) | 1 (1) | 0 | 1 (1) | 6 (10) | 4 (7) | 2 (2)
Pyrexia (General disorders) | 1 (1) | 0 | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1 (1) | 0 | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 | 0 | 0 | 1 (1) | 1 (1) | 0
Blood bilirubin increased (Investigations) | 0 | 1 (1) | 1 (3) | 1 (3) | 2 (2) | 3 (5) | 0
AST increased (Investigations) | 0 | 1 (1) | 0 | 1 (1) | 2 (2) | 1 (2) | 0
ALT increased (Investigations) | 0 | 1 (1) | 0 | 0 | 2 (2) | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 2 (2) | 0 | 1 (1)
Platelet count decreased (Investigations) | 0 | 1 (2) | 0 | 0 | 0 | 0 | 2 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 | 1 (1) | 1 (1) | 1 (1) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 (1) | 0 | 2 (4) | 2 (2) | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 3 (4) | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 (2) | 0 | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 1 (2) | 0 | 3 (6) | 3 (4) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 2 (3) | 0 | 1 (1) | 1 (1) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (2) | 0 | 1 (1) | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 2 (2) | 0 | 0 | 1 (2) | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 (1) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1) | 2 (2) | 0 | 2 (5) | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 (1) | 1 (1) | 1 (3)
Insomnia (Psychiatric disorders) | 1 (1) | 0 | 0 | 1 (1) | 0 | 1 (1) | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 (1) | 2 (3) | 1 (3) | 1 (1) | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 (2) | 1 (1) | 0 | 1 (1) | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 (3) | 0 | 1 (1) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-07-28): https://cdn.clinicaltrials.gov/large-docs/66/NCT04084366/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-12): https://cdn.clinicaltrials.gov/large-docs/66/NCT04084366/SAP_001.pdf